CLINICAL TRIAL: NCT02962960
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 2 Study Characterizing the Pharmacokinetics, Pharmacodynamics, and Safety of Anifrolumab Following Subcutaneous Administration in Adult Systemic Lupus Erythematosus Subjects With Type I Interferon Test High Result and Active Skin Manifestations.
Brief Title: A Study to Characterize the Pharmacokinetics, Pharmacodynamics, and Safety of Anifrolumab in Adult Type I Interferon Test High Systemic Lupus Erythematosus Subject With Active Skin Manifestations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3461C00008
Record Dates: First submitted 2016-09-23; First posted 2016-11-15 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Anifrolumab - Lower dose (Experimental): 1ml, once every second week, one subcutaneous injection as added to stand of care, from week 0 to week 50
  Interventions: Drug: Anifrolumab
- Placebo matching for lower dose of Anifrolumab (Placebo Comparator): 1ml, once every second week, one subcutaneous injection added to stand of care, from week 0 to week 50
  Interventions: Drug: Placebo
- Anifrolumab - Higher dose (Experimental): 2×1ml, once every second week, two subcutaneous injections as added to stand of care, from week 0 to week 50
  Interventions: Drug: Anifrolumab
- Placebo matching for higher dose of Anifrolumab (Placebo Comparator): 2×1ml , once every second week, two subcutaneous injections as added to stand of care, from week 0 to week 50
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anifrolumab — subcutaneous administration every 2 weeks from week 0 to week 50
  Arms: Anifrolumab - Higher dose; Anifrolumab - Lower dose
Drug: Placebo — subcutaneous administration every two weeks from week 0 to week 50
  Arms: Placebo matching for higher dose of Anifrolumab; Placebo matching for lower dose of Anifrolumab

SUMMARY:
This study will be conducted to characterize pharmacokinetics, pharmacodynamics, safety, and tolerability of anifrolumab given via the subcutaneous (SC) route of administration in adult Systemic Lupus Erythematosus (SLE) subjects with a type I Interferon (IFN) test high result and active skin manifestations while receiving Standard of Care (SOC) treatment. In addition, the efficacy of anifrolumab on SLE skin manifestations will be characterized.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 70 years
2. Diagnosis of paediatric or adult SLE for > 24 weeks and fulfilling ≥4 of the 11 American College of Rheumatology (ACR) classification criteria with at least one being:

   * Positive antinuclear antibody (ANA) or
   * Elevated anti-dsDNA antibodies or
   * anti-Smith (anti-Sm) antibodies
3. Interferon high test result
4. Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) activity score ≥ 10
5. Currently receiving at least 1 of the following for treatment of SLE:

   • Oral prednisone or equivalent of ≤40 mg/day for a minimum of 2 weeks prior to signing the Informed Consent Form (ICF) and with stable dose for at least 2 weeks prior to randomization

   • Any of the following medications for at least 12 weeks prior to signing the ICF, and at a stable doses for at least 8 weeks prior to randomization: (i) Azathioprine ≤200 mg/day (ii) Antimalarials (eg, chloroquine, hydroxychloroquine, quinacrine) (iii) Mycophenolate mofetil ≤2 g/day or mycophenolic acid ≤1.44 g/day (iv) Oral, subcutaneous (SC), or intramuscular methotrexate ≤25 mg/week (v) Mizoribine ≤150 mg/day
6. Must not have signs of active or latent tuberculosis (TB).
7. Must not be pregnant or breastfeeding.

Exclusion Criteria:

1. Active severe or unstable neuropsychiatric SLE
2. Active severe SLE-driven renal disease
3. Any severe herpes infection at any time
4. Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or HIV infection.
5. Known history of a primary immunodeficiency (splenectomy, or any underlying condition predisposing for infection
6. Receipt of any investigation product within 4 weeks or 5 half -lives prior to signing of the ICF
7. History of cancer, apart from:

   * Squamous or basal cell carcinoma of the skin if successfully treated.
   * Cervical cancer in situ if successfully treated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (6):
  - Research Site, Thousand Oaks, California
  - Research Site, Orlando, Florida
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Houston, Texas
- Hungary (2):
  - Research Site, Debrecen
  - Research Site, Zalaegerszeg
- Poland (2):
  - Research Site, Bydgoszcz
  - Research Site, Warsaw
- South Korea (4):
  - Research Site, Anyang-si
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Gwangju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruce IN, Nami A, Schwetje E, Pierson ME, Rouse T, Chia YL, Kuruvilla D, Abreu G, Tummala R, Lindholm C. Pharmacokinetics, pharmacodynamics, and safety of subcutaneous anifrolumab in patients with systemic lupus erythematosus, active skin disease, and high type I interferon gene signature: a multicentre, randomised, double-blind, placebo-controlled, phase 2 study. Lancet Rheumatol. 2021 Feb;3(2):e101-e110. doi: 10.1016/S2665-9913(20)30342-8. Epub 2020 Nov 20. PMID 38279367
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3461C00008&attachmentIdentifier=6978de0c-751d-42dc-991c-5a41f7df59f4&fileName=D3461c00008_sap_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants type I Interferon (IFN) test-high Systemic Lupus Erythematosus (SLE) subjects with active skin manifestations while receiving Standard of Care (SOC) treatment were eligible for the study.
Pre-assignment Details: 36 patients were randomized, and all received at least one dose of study treatment.
Groups:
- Placebo Comparator: Pooled placebo comparator to both anifrolumab lower and higher doses, adminstered as either 1ml (1 injection) or 2x1ml (2 injections), once every second week, as added to standar of case, from week 0 to week 50
Period: Overall Study
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator
Started | 14 | 13 | 9
Completed (Subjects who completed study up to Week 52) | 11 | 11 | 9
Not Completed | 3 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes all participants randomized into the study who receive at least one dose of investigational product, according to randomized treatment (modified Intention-To-Treat).
Groups:
- Total: Total of all reporting groups
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator | Total
Number analyzed (Participants) | 14 | 13 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (9.1) | 41.5 (9.2) | 47.8 (14.2) | 44.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 8 | 32
  Male | 2 | 1 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 13 | 9 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 2 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 11 | 9 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration of Anifrolumab in Serum After First Dose
Description: Maximum concentration (Cmax) of anifrolumab is based on sample collected 5 to 8 days after the first dose of strudy treatment.
Time Frame: Week 0
Population: All participants who received anifrolumab and who had at least one quantifiable serum PK observation post first dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose
Number analyzed (Participants) | 13 | 13
mcg/mL | 14.058 (49.8151) | 28.115 (74.4916)

2. Primary Outcome: Steady-state Serum Trough (Predose) Concentration (Ctrough) of Anifrolumab
Description: Steady-state serum through concentration (Ctrough) is based on sample collected at Week 12 prior to dosing of study treatment (predose).
Time Frame: Week 12
Population: All participants who received anifrolumab and who had at least one quantifiable serum PK observation post first dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose
Number analyzed (Participants) | 11 | 11
mcg/mL | 15.618 (81.3595) | 16.926 (9205.6677)

3. Primary Outcome: 21-gene Type 1 IFN Signature Score (Fold-change)
Description: 21-gene type I IFN signature score (fold change) is based on samples collected both at baseline and Week 12 prior to dosing of study treatment. Levels of 21-gene type I IFN pharmacodynamics signature is derived as relative to a pooled normal control.
Time Frame: Week 12
Population: All participants who are 21-gene IFN test high at baseline.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator
Number analyzed (Participants) | 11 | 11 | 9
fold change | 3.2 (3.69) | 3.5 (5.73) | 14.3 (6.68)

4. Primary Outcome: 21-gene Type 1 IFN Neutralization Ratio (Percent Suppression of Fold Change)
Description: 21-gene type I IFN signature score (fold change) is based on samples collected both at baseline and Week 12 prior to dosing of study treatment. For each individual participant and assessment, the level of 21-gene type I IFN pharmacodynamics signature is derived as relative to a pooled normal control, as the median of 100-(((baseline-Week 12)/baseline)*100) for the 21 genes. At a population level, the results are presented as mean the above.
Time Frame: Week 12
Population: All participants who are 21-gene IFN test high at baseline.
Measure: Mean (Standard Deviation); unit: percentage neutralization
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator
Number analyzed (Participants) | 11 | 11 | 9
percentage neutralization | 77.5 (24.16) | 80.5 (36.65) | 15.1 (49.63)

5. Secondary Outcome: Number of Participants With Antidrug Antibody (ADA)
Description: Post-baseline ADA incidence based on the number of participants with Antidrug antibody (ADA)
Time Frame: Baseline to Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator
Number analyzed (Participants) | 14 | 13 | 9
Participants | 1 | 1 | 0

6. Secondary Outcome: Number of Participants With Neutralizing Antibodies (nAb)
Description: Incidence of detectable nAb in post-baseline ADA positive participants.
Time Frame: Baseline to Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator
Number analyzed (Participants) | 1 | 1 | 0
Participants | 0 | 0 | 0

7. Secondary Outcome: Number AEs (Adverse Events) and SAEs (Serious Adverse Events), Including Adverse Events of Special Interest (AESI)
Description: Number of participants with any AEs (Adverse events), any SAEs (serious adverse events), and any adverse events of special interest (AESI) are summarized. More details are reported in the Adverse Events section.
Time Frame: Baseline to Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator
Number analyzed (Participants) | 14 | 13 | 9
Participants
  Any adverse event | 12 | 11 | 7
  Any serious adverse event | 4 | 2 | 0
  Any adverse event of special interest | 5 | 1 | 1

8. Secondary Outcome: Change From Baseline for Vital Signs
Description: Change from baseline for vital signs.
Time Frame: Baseline to Week 60
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo Comparator to Lower Dose: Placebo comparator to anifrolumab lower dose, adminstered as 1ml (1 injection), once every second week, as added to standard of case, from week 0 to week 50
- Placebo Comparator to Higher Dose: Placebo comparator to anifrolumab higher dose, adminstered as 2ml (2 injections), once every second week, as added to standard of case, from week 0 to week 50
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator to Lower Dose | Placebo Comparator to Higher Dose
Number analyzed (Participants) | 14 | 13 | 5 | 4
mmHg
  Systolic Blood Pressure (mmHg) - Week 12: number analyzed (Participants) | 13 | 11 | 5 | 4
  Systolic Blood Pressure (mmHg) - Week 12 | -4.1 (12.08) | 3 (6.63) | -5.8 (13.99) | 7.3 (8.96)
  Systolic Blood Pressure (mmHg) - Week 52: number analyzed (Participants) | 10 | 11 | 5 | 4
  Systolic Blood Pressure (mmHg) - Week 52 | 2.1 (10.96) | -1.7 (12.96) | 3.4 (8.53) | 12.5 (19.36)
  Systolic Blood Pressure (mmHg) - Week 60: number analyzed (Participants) | 9 | 9 | 5 | 4
  Systolic Blood Pressure (mmHg) - Week 60 | 4.1 (19.70) | -2.8 (14.91) | 12.2 (8.61) | 4.5 (7.14)
  Diastolic Blood Pressure (mmHg) - Week 12: number analyzed (Participants) | 13 | 11 | 5 | 4
  Diastolic Blood Pressure (mmHg) - Week 12 | -2.0 (10.02) | 2.4 (6.71) | -3.8 (6.50) | 4.3 (4.35)
  Diastolic Blood Pressure (mmHg) - Week 52: number analyzed (Participants) | 10 | 11 | 5 | 4
  Diastolic Blood Pressure (mmHg) - Week 52 | 0.1 (6.87) | 2.9 (7.54) | -0.4 (7.13) | 6.8 (5.38)
  Diastolic Blood Pressure (mmHg) - Week 60: number analyzed (Participants) | 9 | 9 | 5 | 4
  Diastolic Blood Pressure (mmHg) - Week 60 | 3.6 (12.23) | -0.8 (6.86) | -1.0 (8.22) | 8.8 (6.29)

9. Secondary Outcome: Change From Baseline for Physical Examination
Description: Physical examination is reported as change from baseline in body weight.
Time Frame: Baseline to Week 60
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator to Lower Dose | Placebo Comparator to Higher Dose
Number analyzed (Participants) | 14 | 13 | 5 | 4
kilograms
  Week 12: number analyzed (Participants) | 11 | 10 | 4 | 4
  Week 12 | -1.81 (2.674) | 1.37 (3.113) | 0.7 (1.889) | 0.98 (2.904)
  Week 52: number analyzed (Participants) | 10 | 11 | 5 | 4
  Week 52 | -2.83 (4.683) | 2.52 (6.495) | 0.30 (3.338) | 3.90 (5.608)
  Week 60: number analyzed (Participants) | 8 | 9 | 5 | 4
  Week 60 | -1.81 (3.858) | 2.93 (6.463) | 1.06 (4.020) | 3.60 (5.300)

10. Secondary Outcome: Change From Baseline for 12-lead ECG
Description: The 12-lead ECG measurements were assessed by the investigators, and reported as normal, abnormal (not clinically significant [NCS]), abnormal (clinically significant [CS]), or not done.
Time Frame: Baseline to Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator to Lower Dose | Placebo Comparator to Higher Dose
Number analyzed (Participants) | 14 | 13 | 5 | 4
Participants
  Normal baseline - Normal Week 52 | 7 | 10 | 5 | 3
  Normal baseline - Abnormal (NCS) Week 52 | 1 | 1 | 0 | 0
  Normal baseline - not done Week 52 | 1 | 2 | 0 | 0
  Abnormal (NCS) baseline - Normal Week 52 | 2 | 0 | 0 | 1
  Abnormal (NCS) baseline - Abnormal (NCS) Week 52 | 1 | 0 | 0 | 0
  Abnormal (NCS) baseline - not done Week 52 | 2 | 0 | 0 | 0
  Not done baseline - Normal Week 52 | 0 | 0 | 0 | 0
  Not done baseline - Abnormal (NCS) Week 52 | 0 | 0 | 0 | 0
  Not done baseline - Not done Week 52 | 0 | 0 | 0 | 0
  Normal baseline - Abnormal (CS) Week 52 | 0 | 0 | 0 | 0
  Abnormal (NCS) baseline - Abnormal (CS) Week 52 | 0 | 0 | 0 | 0
  Not done baseline - Abnormal (CS) Week 52 | 0 | 0 | 0 | 0
  Abnormal (CS) baseline - Normal Week 52 | 0 | 0 | 0 | 0
  Abnormal (CS) baseline - Abnormal (CS) Week 52 | 0 | 0 | 0 | 0
  Abnormal (CS) baseline - Not done Week 52 | 0 | 0 | 0 | 0
  Abnormal (CS) baseline - Abnormal (NCS) Week 52 | 0 | 0 | 0 | 0

11. Secondary Outcome: Value of Haemoglobin Blood Test to Detect Change From Baseline
Description: Change from baseline in haemoglobin blood tests are reported.
Time Frame: Baseline to Week 60
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator to Lower Dose | Placebo Comparator to Higher Dose
Number analyzed (Participants) | 14 | 13 | 5 | 4
g/L
  Haemoglobin - Week 12: number analyzed (Participants) | 13 | 11 | 4 | 4
  Haemoglobin - Week 12 | -0.2 (9.07) | 0.7 (7.4) | -0.5 (7.14) | 4.8 (5.91)
  Haemoglobin - Week 52: number analyzed (Participants) | 10 | 10 | 5 | 4
  Haemoglobin - Week 52 | -1.1 (13.92) | 0.1 (11.65) | -4.8 (3.83) | 7 (5.94)
  Haemoglobin - Week 60: number analyzed (Participants) | 8 | 8 | 5 | 4
  Haemoglobin - Week 60 | 0.8 (12.97) | 0 (10.43) | -5.4 (5.68) | 5.8 (6.85)

12. Secondary Outcome: Value of Haematology Blood Tests to Detect Change From Baseline
Description: Change from baseline in haematology blood tests (leucocytes [particle concentration], platelets [particle concentration]) are reported.
Time Frame: Baseline to Week 60
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator to Lower Dose | Placebo Comparator to Higher Dose
Number analyzed (Participants) | 14 | 13 | 5 | 4
10^9/L
  Leucocytes - Week 12: number analyzed (Participants) | 13 | 11 | 4 | 4
  Leucocytes - Week 12 | 0.491 (1.5806) | 3.165 (2.2706) | 0.867 (1.0999) | 1.96 (1.9487)
  Leucocytes - Week 52: number analyzed (Participants) | 10 | 10 | 5 | 4
  Leucocytes - Week 52 | 1.041 (1.5794) | 2.457 (2.3891) | 0.236 (1.0107) | 0.080 (1.4798)
  Leucocytes - Week 60: number analyzed (Participants) | 8 | 8 | 5 | 4
  Leucocytes - Week 60 | -0.012 (1.5489) | 1.474 (1.6490) | 0.776 (2.1779) | 1.23 (1.6687)
  Platelets - Week 12: number analyzed (Participants) | 13 | 11 | 4 | 3
  Platelets - Week 12 | 7.8 (65.28) | 45.2 (67.41) | 10.3 (24.54) | 17.0 (42.58)
  Platelets - Week 52: number analyzed (Participants) | 10 | 9 | 5 | 4
  Platelets - Week 52 | 28.0 (74.28) | 46.1 (74.91) | 6.6 (64.24) | -2.0 (33.85)
  Platelets - Week 60: number analyzed (Participants) | 8 | 8 | 5 | 4
  Platelets - Week 60 | -19.1 (53.48) | 39.0 (60.33) | 24.4 (65.73) | -2.8 (28.43)

13. Secondary Outcome: Value of Protein-creatinine Urinalysis Test to Detect Change From Baseline
Description: Change from baseline in protein-creatinine ratio urinalysis tests are reported.
Time Frame: Baseline to Week 60
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: g/g
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator to Lower Dose | Placebo Comparator to Higher Dose
Number analyzed (Participants) | 14 | 13 | 5 | 4
g/g
  Protein/Creatinine - Week 12: number analyzed (Participants) | 13 | 11 | 4 | 3
  Protein/Creatinine - Week 12 | 1.37029 (5.186672) | -0.13007 (1.123807) | -0.03056 (0.056701) | 0.32764 (0.337631)
  Protein/Creatinine - Week 52: number analyzed (Participants) | 10 | 10 | 5 | 4
  Protein/Creatinine - Week 52 | 0.03756 (0.135157) | -0.00465 (0.183327) | -0.00781 (0.047671) | 0.080930 (1.581772)
  Protein/Creatinine - Week 60: number analyzed (Participants) | 9 | 8 | 5 | 4
  Protein/Creatinine - Week 60 | 0.02578 (0.119862) | -0.28836 (1.185347) | -0.03501 (0.061888) | 0.46178 (0.899886)

14. Secondary Outcome: Value of Total Protein Urinalysis Test to Detect Change From Baseline
Description: Change from baseline in total protein urinalysis tests are reported.
Time Frame: Baseline to Week 60
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator to Lower Dose | Placebo Comparator to Higher Dose
Number analyzed (Participants) | 14 | 13 | 5 | 4
g/L
  Protein, Total - Week 12: number analyzed (Participants) | 13 | 11 | 4 | 3
  Protein, Total - Week 12 | 0.7669 (2.71221) | -0.0744 (0.76445) | 0 (0) | 0.3443 (0.34301)
  Protein, Total - Week 52: number analyzed (Participants) | 10 | 10 | 5 | 4
  Protein, Total - Week 52 | -0.0029 (0.08124) | -0.0011 (0.33468) | 0 (0) | 0.1143 (0.24476)
  Protein, Total - Week 60: number analyzed (Participants) | 9 | 9 | 5 | 4
  Protein, Total - Week 60 | 0.1151 (0.12514) | -0.1790 (0.83066) | 0.003 (0.00671) | 0.3975 (0.82602)

15. Secondary Outcome: Value of Clinical Chemistry Blood Tests to Detect Change From Baseline (Serum)
Description: Change from baseline in clinical chemistry blood tests (Alanine Aminotransferase, Aspartate Aminotransferase) are reported.
Time Frame: Baseline to Week 60
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator to Lower Dose | Placebo Comparator to Higher Dose
Number analyzed (Participants) | 14 | 13 | 5 | 4
ukat/L
  Alanine Aminotransferase - Week 12: number analyzed (Participants) | 13 | 10 | 4 | 3
  Alanine Aminotransferase - Week 12 | 0.00769 (0.147479) | -0.13003 (0.431764) | -0.05418 (0.045905) | 0.02501 (0.134397)
  Alanine Aminotransferase - Week 52: number analyzed (Participants) | 10 | 11 | 5 | 4
  Alanine Aminotransferase - Week 52 | -0.06335 (0.119642) | -0.05607 (0.556152) | -0.06335 (0.047735) | 0.04167 (0.169182)
  Alanine Aminotransferase - Week 60: number analyzed (Participants) | 9 | 9 | 5 | 4
  Alanine Aminotransferase - Week 60 | -0.01297 (0.043131) | 0.09446 (0.365981) | -0.04334 (0.032495) | -0.01667 (0.18127)
  Aspartate Aminotransferase - Week 12: number analyzed (Participants) | 13 | 10 | 4 | 4
  Aspartate Aminotransferase - Week 12 | -0.01154 (0.065765) | -0.10502 (0.169099) | 0.00417 (0.059911) | 0.03334 (0.105430)
  Aspartate Aminotransferase - Week 52: number analyzed (Participants) | 10 | 11 | 5 | 4
  Aspartate Aminotransferase - Week 52 | -0.04834 (0.066424) | -0.05304 (0.196369) | 0.00333 (0.090847) | 0.09169 (0.100482)
  Aspartate Aminotransferase - Week 60: number analyzed (Participants) | 9 | 9 | 5 | 4
  Aspartate Aminotransferase - Week 60 | -0.01111 (0.058937) | 0.04816 (0.123752) | 0 (0.050010) | -0.02501 (0.099555)

16. Secondary Outcome: Value of Creatinine Clinical Chemistry Blood Tests to Detect Change From Baseline (Serum)
Description: Change from baseline in clinical creatinine chemistry blood tests (serum) are reported.
Time Frame: Baseline to Week 60
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator to Lower Dose | Placebo Comparator to Higher Dose
Number analyzed (Participants) | 14 | 13 | 5 | 4
umol/L
  Creatinine - Week 12: number analyzed (Participants) | 13 | 10 | 4 | 4
  Creatinine - Week 12 | 4.385 (8.5799) | -3.6 (11.2467) | 5.5 (6.3509) | 5.25 (9.8446)
  Creatinine - Week 52: number analyzed (Participants) | 10 | 11 | 5 | 4
  Creatinine - Week 52 | 12.2 (33.2597) | -7.273 (19.5862) | 0.2 (13.9714) | 2.5 (5.5076)
  Creatinine - Week 60: number analyzed (Participants) | 9 | 9 | 5 | 4
  Creatinine - Week 60 | 7.316 (8.7449) | -5.556 (12.8463) | 5.0 (10.4163) | 6.5 (12.5033)

17. Secondary Outcome: Value of Inflammatory Marker Panel Blood Tests to Detect Change From Baseline
Description: Change from baseline in the Erythrocyte Sedimentation Rate (ESR) inflammatory marker is reported.
Time Frame: Baseline to Week 60
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator
Number analyzed (Participants) | 14 | 13 | 9
mm
  ESR - Week 12: number analyzed (Participants) | 12 | 11 | 8
  ESR - Week 12 | -3.0 (20.37) | -7.2 (15.46) | -11.9 (15.36)
  ESR - Week 52: number analyzed (Participants) | 9 | 10 | 9
  ESR - Week 52 | 5.6 (25.58) | -6.7 (12.25) | -16.0 (10.95)
  ESR - Week 60: number analyzed (Participants) | 7 | 9 | 9
  ESR - Week 60 | 14.6 (38.77) | -1.0 (21.84) | 2.2 (22.48)

18. Secondary Outcome: Value of Autoantibody Blood Panel Blood Tests to Detect Change From Baseline
Description: Change from baseline in Anti-Double Stranded DNA IgG (anti-dsDNA) is reported.
Time Frame: Baseline to Week 60
Population: Includes all participants randomized into the study who receive at least one dose of investigational product, according to randomized treatment (modified Intention-To-Treat). Only participants with abnormal baseline values are included in this analysis.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator to Lower Dose | Placebo Comparator to Higher Dose
Number analyzed (Participants) | 9 | 8 | 3 | 3
IU/mL
  anti-dsDNA - Week 12: number analyzed (Participants) | 9 | 7 | 2 | 3
  anti-dsDNA - Week 12 | -42.09 (256.228) | -84.97 (231.489) | -37.0 (19.799) | -97.33 (151.596)
  anti-dsDNA - Week 52: number analyzed (Participants) | 7 | 6 | 3 | 3
  anti-dsDNA - Week 52 | -99.04 (288.183) | 8.70 (27.308) | -13.0 (50.229) | -76.87 (127.433)
  anti-dsDNA - Week 60: number analyzed (Participants) | 6 | 6 | 3 | 3
  anti-dsDNA - Week 60 | 52.67 (144.220) | 16.53 (30.528) | -21.33 (54.921) | -76.73 (141.525)

19. Secondary Outcome: Number of Participants With Positive Hepatitis B Core Antibody Post-baseline.
Description: Change from screening in Hepatitis B core antibody was monitored during the study for participants tested positive at screening.
Time Frame: Baseline to Week 60
Population: Includes all participants randomized into the study who receive at least one dose of investigational product, according to randomized treatment (modified Intention-To-Treat). No participants were positive for Hepatitis B at screening, therefore no participants were tested post-baseline.
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator to Lower Dose | Placebo Comparator to Higher Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: An unfavorable change in the health of a participant, including abnormal laboratory findings, that happens during the clinical study (from and including the day of first dose of investigational product, up to, and including, the date of last dose of investigational product pluts 14 days). This change may or may not be caused by the treatment being studied.
Arm/Group | Anifrolumab - Lower Dose | Anifrolumab - Higher Dose | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/9
Serious Adverse Events (participants affected / at risk) | 4/14 | 2/13 | 0/9
Other Adverse Events (participants affected / at risk) | 12/14 | 11/13 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anifrolumab - Lower Dose (N=14) | Anifrolumab - Higher Dose (N=13) | Placebo Comparator (N=9)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis Media Acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Lupus Nephritis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anifrolumab - Lower Dose (N=14) | Anifrolumab - Higher Dose (N=13) | Placebo Comparator (N=9)
Abscess Limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acute Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 3 (5) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (9) | 1 (1) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial Cyst (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal Septum Perforation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia Oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Anembryonic Gestation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Endometrial Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Face Oedema (General disorders) | 0 (0) | 1 (2) | 0 (0)
Feeling Hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mycobacterium Tuberculosis Complex Test Positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-09-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT02962960/Prot_002.pdf
  • Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT02962960/SAP_001.pdf